CLINICAL TRIAL: NCT04711694
Title: Early Mindfulness-based Intrevention for Anxious Adolescents: a fMRI Randomized Controlled Trial
Brief Title: Mindfulness-Based Intervention for Adolescents
Acronym: Mindfulteen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: Leenards Foundation (Unknown); University of Lausanne (Other); Swiss National Centre Competence in Research - Synapsy (Unknown)
Responsible Party: Principal Investigator, Camille Nemitz Piguet, Postdoc at centre Neurospin Paris, University of Geneva, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-017731
Record Dates: First submitted 2019-05-16; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Anxiety; Adolescent Behavior; Stress
Keywords: Adolescent; Mindfulness; Anxiety; Stress; Teenager; MRI; Intervention
MeSH Terms: conditions — Anxiety Disorders; Adolescent Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants cannot be blinded to MBI time (early vs late). Outcome assessors are blind to intervention group. One of the two mindfulness instructors is not blind, as she works as clinical research coordinator. However, MBI are always held by both instructors together and the groups are mixed between early and late intervention allocated participants, diminishing the impact of the lack of blinding of one instructor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Mindfulness Intervention (Experimental): The Early MBI group partake on the mindfulness intervention after first outcome assessment.
  Interventions: Behavioral: Minfulness-based Intervention
- Late Mindfulness Intervention (Placebo Comparator): The Late MBI group partake on the mindfulness intervention after the second outcome assessment.
  This groups is the control group for the Early MBI group.
  After the second assessment, this group engage on the same intervention as the early group.
  Interventions: Behavioral: Minfulness-based Intervention

INTERVENTIONS:
Behavioral: Minfulness-based Intervention — The proposed MBI is an adaptation from the Mindfulness Based Stress Reduction (MBSR) and Mindfulness based Cognitive Therapy (MBCT) programs to youth. This MBI consists of a total of twelve 90 minutes long sessions, the first 8 being the intervention per se and the last 4 a proposition to the transition to regular practice and a chance to better integrate mindfulness in daily life.
  A theme regarding mindfulness is addressed in each session, through meditation practices and exercises. Between sessions, participants are invited to practice at home, using an application designed for this study (the MindApp), where participants can find the recorded practices. Investigators have access to participants' use of the meditation recordings and expect that these data will provide a more objective measure of the amount of home practice.

SUMMARY:
The Mindfulteen Study is a 3-year long longitudinal cohort study with a nested randomized controlled trial, integrating neuroimaging, biological and clinical outcomes, and designed to evaluate the impact of a mindfulness-based intervention (MBI) on young adolescents.

Young adolescents between 13 and 15 years with no history of current mental health disorder (with the exception for anxiety symptoms) or of psychotherapy are included and randomized to either early or late intervention (i.e. waiting list or control group), after being stratified between low or high anxiety group based on State and Trait Anxiety Inventory (STAI-T) score. Participants on the control group participate on MBI after completing the second assessment. The intervention is an 8-week long MBI adapted to adolescents. Primary outcomes are based on neuroimaging (structural and functional MRI) and secondary outcomes are clinical (self-reported questionnaires covering mostly emotion and stress reactivity and trait mindfulness) and biological (cortisol, inflammation markers and redox markers). Assessments are performed at baseline, immediately after intervention or waiting time and after 18 months of intervention.

DETAILED DESCRIPTION:
Promotion of mental health is a major concern worldwide, particularly among young population as major psychiatric diseases can have their onset during adolescence and young adulthood. During adolescence, there is growing evidence that "at-risk" states for mental disorders, as high stress reactivity for example, can be identified prior to clinical symptoms, and that early interventions can have a major impact preventing the further development of full-blown mental illness.

In the last two decades, given a growing interest for non-pharmacological approaches to improve mental and physical health, mindfulness-based interventions (MBI) have received serious attention. After the initial applications on chronic pain, stress reduction and prevention of depressive relapses, MBIs are now widely implemented among clinical and non-clinical populations.

Therefore, investigators aim to better understand the modifications of brain circuits involved in the emergence of stress related disorders and the impact of a MBI on those circuits. Hence, a translational project was designed, integrating neuroimaging, biological and clinical outcomes of stress reactivity to evaluate the impact of a MBI on adolescents.

The Mindfulteen Study is a 3-year longitudinal cohort study with a nested randomized controlled trial. The randomized controlled trial part of the study was designed to assess the clinical effect of MBI on adolescents, comparing to a control group. Therefore, after inclusion participants are electronically randomized between either early intervention group or late intervention group (i.e., waiting list or control group). Participants allocated in the late intervention group engage in MBI after the waiting period, providing data also for the longitudinal cohort part of the study and therefore increasing the data available for before and after comparison. The long-term effect of MBI will be assessed after 18 months of intervention.

Before randomization, participants are stratified according to their score on the trait questionnaire of the State Trait Anxiety Inventory (STAI) as low anxiety group (≤ 31) or high anxiety group (>31).

Assessments are performed before intervention, immediately after intervention or waiting period and in 18 months. For the late intervention group, an additional assessment is performed immediately after the intervention.

The overall objective of the Mindfulteen Study is to assess the immediate and long-term effect of an MBI on reactivity to stress and anxiety, in a non-clinical sample of young adolescents from the general population. Underlying psychological and biological changes are assessed using a multimodal brain MRI protocol, blood and hair sampling, as well as physiological measurements of stress.

The primary aim is to characterize brain functional modifications in cortico-limbic and cortico-striatal-thalamic circuits (functional MRI data) and their underlying neuroanatomical changes (analysis of structural, spectroscopy and diffusion MRI data) in adolescents exposed to MBI, comparing adolescents with high anxiety and low anxiety levels.

Secondary aims include the effects of MBI on self-reported levels of anxiety, emotion regulation strategies (clinical scores) and physiological markers of hypothalamic-pituitary-adrenal axis (hair cortisol), as well as biological markers of oxidative stress and inflammation (blood sampling).

ELIGIBILITY:
Inclusion Criteria:

* Age 13 to 15 year-old
* Interest in participating in a mindfulness based intervention
* Francophone
* Have access to internet and a to a compatible device (smartphone or tablet) every day to run the study's application
* Availability for the study duration
* Consent documented by signature and support from the legal representatives as documented by a signature
* Informed Consent as documented by a signature

Exclusion Criteria:

* History of chronic somatic disease or clinically significant medical condition (e.g., asthma, diabetes, renal failure, hepatic dysfunction, etc.)
* History of neurologic or major psychiatric disease (except for an anxious disorder without comorbidity and a history of major depressive episode resolved for at least 6 months).
* History of psychotherapy in the past 6 months
* History of regular meditation practice
* Women who are pregnant or breast feeding
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to participate in group sessions,
* Previous enrolment into the current study
* Inability to undergo study's procedures (IRM and blood sample collection)

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Brain activity in stress-related networks at functional MRI | At baseline, immediately after intervention, 18 months after intervention
  Change of the fronto-limbic circuit recovery after a social laboratory stress using the Montreal Imaging Stress Task (MIST)
Brain gray matter at structural MRI | At baseline, immediately after intervention, 18 months after intervention
  Change on gray matter volume in prefrontal areas
Brain connectivity at functional MRI | Before and after intervention
  Change in structural connectivity measures between prefrontal and limbic areas after intervention
Brain cortical thickness at structural MRI | At baseline, immediately after intervention, 18 months after intervention
  Cortical thickness in prefrontal areas

SECONDARY OUTCOMES:
Level of anxiety | At baseline, immediately after intervention, 18 months after intervention
  Change of the level of anxiety measured by the State and Trait Anxiety Inventory. Minimum score 20, maximum score 60. Higher score means a worse outcome (higher anxiety).
Level of emotional awareness | At baseline, immediately after intervention, 18 months after intervention
  Change on the baseline Emotion Awareness Questionnaire score after intervention. Minimum score 0, maximum score 40. Higher score means a better outcome.
Level of emotional regulation | At baseline, immediately after intervention, 18 months after intervention
  Change on the baseline Emotion Regulation Questionnaire score after intervention. Minimum score 6, maximum score 30. Higher score means a better outcome.
Level of inflammation | At baseline, immediately after intervention, 18 months after intervention
  Change on baseline innate immunity-related proteins after intervetion, measured in pg/ml.
Level redox system activity | At baseline, immediately after intervention, 18 months after intervention
  Change on the baseline activity of plasma glutathion and metabolites after intervention, measured in mMol/L-
Hair cortisol level | At baseline, immediately after intervention, 18 months after intervention
  Change on the baseline hair cortisol measure after intervention, measured in pg/mg.
Heart rate variability | At baseline, immediately after intervention, 18 months after intervention
  Change on baseline herat rate variability after intervetion.
Level of redox system activity | At baseline, immediately after intervention, 18 months after intervention
  Change on baseline activity of enzimes involved in glutathion metabolism after intervention, measured in U/gHb

CONTACTS AND LOCATIONS:
Overall Officials: Camille Piguet, Physician, Principal Investigator — Geneva University
Locations (1):
- Geneva University, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piguet C, Celen Z, Meuleman B, Schilliger Z, Magnus Smith M, Mendola E, Pham E, Jouabli S, Ivanova V, Murray RJ, Klauser P, Merglen A. Impact of a Mindfulness-Based Intervention on Symptoms and Emotion Regulation Strategies in Young Adolescents From the General Population: A Randomized Controlled Trial. Depress Anxiety. 2025 Jun 10;2025:2679049. doi: 10.1155/da/2679049. eCollection 2025. PMID 40529112